CLINICAL TRIAL: NCT00785473
Title: Can Vitamin D Supplementation Prevent Bone Loss in Persons With MS? A Randomised, Placebo-controlled, Single-centre Study
Brief Title: Can Vitamin D Supplementation Prevent Bone Loss in Persons With Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSvitD1; EudraCT 2006-00427-11
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Sclerosis, Osteoporosis
MeSH Terms: conditions — Multiple Sclerosis; Osteoporosis | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): cholecalciferol, calcium carbonate
  Interventions: Dietary Supplement: cholecalciferol; Dietary Supplement: calcium carbonate
- 2 (Placebo Comparator): capsules not containing cholecalciferol, otherwise identical to Active comparator; calcium carbonate
  Interventions: Dietary Supplement: calcium carbonate

INTERVENTIONS:
Dietary Supplement: cholecalciferol — cholecalciferol capsules, 20,000 IU weekly for 2 years and calcium carbonate 500 mg daily
  Other Names: Dekristol, Weifa-kalsium
  Arms: 1
Dietary Supplement: calcium carbonate — calcium carbonate 500 mg daily for 2 years
  Other Names: Weifa-kalsium

SUMMARY:
Several studies have shown that bone mineral density (BMD) at the femoral neck decreases with increasing physical handicap (EDSS-score) in MS patients. Possible explanations are less weightbearing exercise or less UV-exposure resulting in reduced vitamin D generation in the skin. Prevention of osteoporosis is a high priority, because treatment of the established disease remains sub-optimal.

We have designed a double-blind randomised controlled trial of two years' duration including 90-100 persons with MS age 18-50 to assess whether supplementation with vitamin D, given as a weekly dose of 20,000 IU cholecalciferol, can prevent bone loss.

The primary objective of this study is to determine changes in BMD over the 2 year study period comparing treatment and placebo groups.

The most important secondary objective is to determine cytokine profiles in blood samples. We will also assess parameters related to vitamin D status and physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* EDSS < 4.0 (able to walk without rest some 500 m)
* Women have to be premenopausal
* MS according to the McDonald criteria; prepared and considered able to follow the protocol; using appropriate contraceptive methods (women of childbearing potential)
* Having given written informed consent.

Exclusion Criteria:

* Pregnancy or unwillingness to use contraception; alcohol or drug abuse
* Use of glucocorticoid treatment other than intravenous methylprednisolone for treatment of relapses
* Known allergy to cholecalciferol or arachis oil (peanuts)
* Therapy with digitalis, calcitonin, active vitamin D3 analogues, fluoride, or bisphosphonates during the previous 12 months
* Any condition predisposing to hypercalcaemia
* Nephrolithiasis or renal insufficiency
* Presence of primary hyperparathyroidism, hyperthyroidism, or hypothyroidism in the year before the study began; a history of nephrolithiasis during the previous five years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Changes in BMD over the 2 year study period comparing treatment and placebo groups | 2 years

SECONDARY OUTCOMES:
Cytokine expression following vitamin D supplementation | 2 years
Contribution of vitamin D from different sources (generation in the skin, diet and supplements) to serum 25(OH) vitamin D (vitamin D status) | 2 years
Changes in parameters of lower extremity function over the 2 year study period | 2 years
The number of relapses, the time to first relapse, the number of relapse-free patients | 2 years
The number of patients without progression of disability judged by EDSS and | 2 years
Reported infections | 2 years
Ratings on a fatigue scale | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Margitta T Kampman, MD, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Holmoy T, Lindstrom JC, Eriksen EF, Steffensen LH, Kampman MT. High dose vitamin D supplementation does not affect biochemical bone markers in multiple sclerosis - a randomized controlled trial. BMC Neurol. 2017 Apr 4;17(1):67. doi: 10.1186/s12883-017-0851-0. PMID 28376767
- [Derived] Rosjo E, Lossius A, Abdelmagid N, Lindstrom JC, Kampman MT, Jorgensen L, Sundstrom P, Olsson T, Steffensen LH, Torkildsen O, Holmoy T. Effect of high-dose vitamin D3 supplementation on antibody responses against Epstein-Barr virus in relapsing-remitting multiple sclerosis. Mult Scler. 2017 Mar;23(3):395-402. doi: 10.1177/1352458516654310. Epub 2016 Jul 11. PMID 27325604
- [Derived] Kampman MT, Steffensen LH, Mellgren SI, Jorgensen L. Effect of vitamin D3 supplementation on relapses, disease progression, and measures of function in persons with multiple sclerosis: exploratory outcomes from a double-blind randomised controlled trial. Mult Scler. 2012 Aug;18(8):1144-51. doi: 10.1177/1352458511434607. Epub 2012 Feb 21. PMID 22354743
- [Derived] Steffensen LH, Jorgensen L, Straume B, Mellgren SI, Kampman MT. Can vitamin D supplementation prevent bone loss in persons with MS? A placebo-controlled trial. J Neurol. 2011 Sep;258(9):1624-31. doi: 10.1007/s00415-011-5980-6. Epub 2011 Mar 13. PMID 21400196